CLINICAL TRIAL: NCT07079215
Title: A Single Center, Double-Blind, Randomized, Sham-Controlled, Parallel Design, Exploratory Clinical Trial to Evaluate the Safety and Efficacy of a Medical Device for the Treatment of Opioid Withdrawal Symptoms
Brief Title: Evaluation of a Physical Device for Medical Use (ADTPM 1) for Opioid Withdrawal Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nu Eyne Co., Ltd. (Industry)
Collaborators: C&R Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE_ADT_001
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Opioid Withdrawal (Disorder); Opioid Use Disorder
Keywords: OUD
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group (Active Stimulation, n=12):
  Participants in this group will use the physical device for medical use (ADTPM 1) applied to the auricular region (ear and surrounding area) for 60 minutes (±10 minutes) per session, at least once daily and a minimum of 7 times per week, over a 4-week treatment period. Additional sessions may be conducted if participants require further relief of withdrawal symptoms. All assessments and permitted concomitant treatments will be administered in accordance with the study protocol.
  Interventions: Device: Neurostimulation
- Control Group (Sham Comparator): Control Group (Sham Stimulation, n=12):
  Participants in this group will use a sham stimulation device that does not deliver active stimulation. The sham device will be applied under the same schedule and conditions-60 minutes (±10 minutes) per session, at least once daily and 7 times per week for 4 weeks. All assessments and permitted concomitant treatments will be identical to those in the active stimulation group.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Neurostimulation — Participants in this group will use the physical device for medical use (ADTPM 1) applied to the auricular region (ear and surrounding area) for 60 minutes (±10 minutes) per session, at least once daily and a minimum of 7 times per week, over a 4-week treatment period. Additional sessions may be conducted if participants require further relief of withdrawal symptoms. All assessments and permitted concomitant treatments will be administered in accordance with the study protocol.
  Other Names: ADTPM 1
  Arms: Experimental Group
Device: Sham stimulation — Control Group (Sham Stimulation, n=12):
  Participants in this group will use a sham stimulation device that does not deliver active stimulation. The sham device will be applied under the same schedule and conditions-60 minutes (±10 minutes) per session, at least once daily and 7 times per week for 4 weeks. All assessments and permitted concomitant treatments will be identical to those in the active stimulation group.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the safety and efficacy of a physical device for medical use (ADTPM 1) applied to opioid withdrawal symptoms.

DETAILED DESCRIPTION:
This study is a single-center, double-blind, randomized, sham-controlled, parallel-design exploratory clinical trial to evaluate the safety and efficacy of a physical device for medical use (ADTPM 1) in adults with opioid withdrawal symptoms. Eligible participants will be randomized to receive either active stimulation or sham stimulation applied to the auricular region daily for 60 minutes over a 4-week period. The primary objective is to assess the incidence of treatment-emergent adverse events. Secondary objectives include evaluating changes in opioid withdrawal severity, craving, pain, heart rate, depressive symptoms, anxiety, insomnia, somatic symptoms, and DSM-5 criteria for opioid use disorder over time.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 19 to 80 years
2. Participants currently dependent on opioids, whether prescribed or non-prescribed
3. Participants who meet the criteria for opioid use disorder (OUD) according to DSM-5
4. Participants with a Clinical Opiate Withdrawal Scale (COWS) score of 5 or higher
5. Participants with a Numeric Rating Scale (NRS) pain score of less than 6
6. Participants who have voluntarily decided to participate in the study and have provided written informed consent
7. Participants who are willing to comply with the study protocol

Exclusion Criteria:

1. Participants with any current uncontrolled or clinically significant medical condition
2. Participants with a history of seizures or epilepsy
3. Participants with a history of neurological disorders or traumatic brain injury
4. Participants who have used long-acting opioids, such as methadone or buprenorphine, continuously for more than 5 days prior to screening
5. Participants who have used methadone within 30 days prior to screening
6. Participants who have used buprenorphine within 7 days prior to screening
7. Participants with physiological dependence on alcohol or drugs other than opioids, tobacco, or marijuana
8. Participants diagnosed with a major psychiatric disorder (psychosis, schizophrenia, or bipolar disorder)
9. Participants who are currently hospitalized due to a recent suicide attempt or who are persistently expressing suicidal intent
10. Participants with implanted devices such as a pacemaker, cochlear implant, or neurostimulator.
11. Participants with abnormal ear anatomy or ear infections
12. Participants diagnosed with renal or hepatic failure
13. Participants who are currently undergoing chemotherapy (Exception: Participation may be allowed if the investigator determines that participation poses no medical safety concerns for the participant)
14. Participants who are currently engaged in high-risk occupations (e.g., transportation workers, crane operators, heavy machinery operators, individuals working with sharp objects, or those requiring a high level of cognitive functioning)
15. Participants with implanted metal or electronic devices in the head or neck area, including deep brain stimulators or pacemakers, as specified in the product precautions and contraindications (dental implants are exempt)
16. Participants with cognitive impairment due to neurodevelopmental disorders (e.g., intellectual disability, developmental disorders, autism spectrum disorder) or neurodegenerative disorders (e.g., Alzheimer's disease, vascular dementia) that would make it difficult to undergo treatment with the investigational medical device
17. Participants who are pregnant or breastfeeding
18. Female participants of childbearing potential who do not agree to abstain from sexual intercourse or to use medically accepted contraception* during the study period.

    *Medically accepted methods of contraception include: condoms, consistent oral contraceptive use (≥3 months use), injectables or implantable contraceptives, or intrauterine devices (IUDs).
19. Participants who are currently participating in another clinical trial or who have participated in another clinical trial within 30 days prior to screening
20. Participants who, in the opinion of the investigator, are deemed inappropriate for participation due to ethical concerns or potential impacts on study outcomes

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | [Time Frame: Baseline to Week 4]
  The primary outcome is the incidence and severity of treatment-emergent adverse events (TEAEs) occurring from the first device application through the end of the 4-week treatment period. TEAEs include, but are not limited to, mild adverse events such as dizziness, somnolence, skin irritation, and headache. Safety will be assessed by monitoring vital signs, conducting physical examinations, and recording adverse events throughout the study period.

SECONDARY OUTCOMES:
Change in Clinical Opiate Withdrawal Scale (COWS) Scores | [Time Frame: Baseline, 1 Hour, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change from baseline in COWS scores to assess the severity of opioid withdrawal symptoms over time. Higher scores indicate more severe withdrawal symptoms.
Change in Subjective Opiate Withdrawal Scale (SOWS) Scores | [Time Frame: Baseline, 1 Hour, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change from baseline in SOWS scores to evaluate patient-reported withdrawal symptoms. Higher scores indicate more severe withdrawal symptoms.
Change in Opioid Craving Visual Analogue Scale (OC-VAS) | [Time Frame: Baseline, 1 Hour, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in opioid craving levels measured by a visual analogue scale. Higher scores indicate more severe craving.
Change in Heart Rate | [Time Frame: Baseline, 1 Hour, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in resting heart rate from baseline to assess physiological responses related to withdrawal. Higher heart rate may reflect increased autonomic arousal associated with withdrawal.
Change in Numerical Rating Scale (NRS) | [Time Frame: Baseline, 1 Hour, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in self-reported pain severity measured by the NRS. Higher scores indicate greater pain intensity.
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Scores | [Time Frame: Baseline, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in depressive symptom severity from baseline. Higher scores indicate more severe depressive symptoms.
Change in Generalized Anxiety Disorder-7 (GAD-7) Scores | [Time Frame: Baseline, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in anxiety symptom severity from baseline. Higher scores indicate more severe anxiety symptoms.
Change in Insomnia Severity Index-Korean (ISI-K) Scores | [Time Frame: Baseline, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in insomnia symptoms assessed by ISI-K. Higher scores indicate more severe insomnia symptoms.
Change in Patient Health Questionnaire-15 (PHQ-15) Scores | [Time Frame: Baseline, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in somatic symptom severity over the treatment period. Higher scores indicate more severe somatic symptoms.
Change in DSM-5 Criteria for Opioid Use Disorder | [Time Frame: Baseline, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in diagnostic status of opioid use disorder as defined by DSM-5. Meeting more criteria indicates greater disorder severity
Change in Opioid Craving Scale (OCS-3) Scores | [Time Frame: Baseline, Day 2, Week 1, Week 2, Week 3, Week 4]
  Change in opioid craving symptoms measured by OCS-3. Higher scores indicate more severe craving.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided